CLINICAL TRIAL: NCT04734340
Title: The Study of EIT-guided Ventilation Strategy on ARDS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EIT-RCT
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: ARDS; Pulmonary Perfusion
Keywords: EIT; ARDS; pulmonary perfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT-guided group (Experimental): Treatment based on EIT
  Interventions: Procedure: EIT-guided PEEP setting
- Control group (Placebo Comparator): Treatment based on ARDS-net Peep setting
  Interventions: Procedure: ARDS-net PEEP setting

INTERVENTIONS:
Procedure: EIT-guided PEEP setting — Ventilator parameter setting by EIT
  Arms: EIT-guided group
Procedure: ARDS-net PEEP setting — Ventilator parameter setting according to ARDS-net table
  Arms: Control group

SUMMARY:
This study is a clinical randomized controlled study.The objective of this study is to compare the prognosis of patients with ARDS between eit-v / q-oriented individualized ventilation strategy and traditional lung protection ventilation strategy, and to establish the demonstration application of eit-v / q-oriented ventilation strategy in ARDS

ELIGIBILITY:
Inclusion Criteria:

1. According to ARDS Berlin standard, ARDS, PaO2 / FiO2 < 200mmhg, peep > 5cmh2o;
2. According to clinical judgment, lung recruitment therapy is needed due to hypoxemia;
3. The subjects or their families signed informed consent.
4. Admission to ICU was less than 72 hours;
5. The estimated duration of mechanical ventilation was more than or equal to 48 hours;
6. Age ≥ 18 years old and ≤ 80 years old;

Exclusion Criteria:

1. The patients with heart implants could not be monitored by EIT;
2. Patients or their families refused to participate in the study;
3. Hypernatremia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
ventilation free days | 1 Day

SECONDARY OUTCOMES:
28-day mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No